CLINICAL TRIAL: NCT03764670
Title: The Influence of Genetic and Clinical Factors on Clinical Outcomes of Kidney Transplant Patients With Tacrolimus Based Immunosuppression
Brief Title: Genetic Factors on Outcomes of Kidney Transplant Patients With Tacrolimus-based Therapy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201809018RINB
Record Dates: First submitted 2018-11-15; First posted 2018-12-05 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2020-09

CONDITIONS: Kidney Transplantation
Keywords: tacrolimus; clinical outcomes; genetic polymorphism; clinical factors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify the influence of genetic and clinical factors on the clinical outcomes of kidney transplant patients with tacrolimus (TAC) based immunosuppression in Taiwan.

DETAILED DESCRIPTION:
Tacrolimus (TAC) is the most important immunosuppressants for maintenance therapy after kidney transplantation. Many genetic and clinical factors had been found to have effect on TAC pharmacokinetics (PK). Whether these factors affect clinical outcomes is still controversial.

In this retrospective study, investigators will review records of kidney transplant patients with TAC based immunosuppression recruited from a previous study (IRB approval number: 201512005RINC) to understand the influence of clinical and genetic factors on their 3-years clinical outcomes, including biopsy-proven acute rejection, patient survival, graft survival and safety issues of kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplantation
2. 20-65 years old
3. Receiving tacrolimus-based immunosuppressants
4. Were recruited in a previous trial

Exclusion Criteria:

1. Human immunodeficiency virus-positive status
2. Retransplantation or multiorgan transplantation
3. Non-Asian

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients who underwent transplantation at National Taiwan University Hospital, and received tacrolimus based immunosupression
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Acute rejection | Within the first 1 year post-transplantation
  The incidence of acute rejection within the first 1 year post-transplantation, estimated with Kaplan-Meier survival analysis
Graft survival | From post-transplantation to Dec 31, 2017
  The incidence of graft loss during the follow-up time, estimated with Kaplan-Meier survival analysis

SECONDARY OUTCOMES:
Patient survival | From post-transplantation to Dec 31, 2017
  The incidence of death during the follow-up time (number of events or frequency)
Kidney function measured by estimated glomerular filtration rate (eGFR) | From post-transplantation to Dec 31, 2017
  Kidney function during the follow-up time measured by eGFR (MDRD 4-variable equation, in mL/min/1.73 m^2).
Incidence of adverse events, including post-transplant diabetes mellitus, deterioration of liver function, cancer, infection and hyperlipidemia | From post-transplantation to Dec 31, 2017
  The incidence of infection and cancer in number of events or frequency in percentage.
  The change of liver function : measured by aspartate aminotransferase (AST in U/L), alanine aminotransferase (ALT in U/L), and total bilirubin in mg/dL.
  Hyperlipidemia: identified by diagnosis and the use of lipid-lowering agents, with follow-up of LDL in mg/dL, HDL in mg/dL, and total cholesterol in mg/dL.
  Post-transplant diabetes mellitus: identified by diagnosis and the use of antihyperglycemic agents, with follow-up of hemoglobin A1c in percentage and blood glucose in mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Kun Tsai, Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan